CLINICAL TRIAL: NCT05003921
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intrathecal Injection for the Treatment of Amyotrophic Lateral Sclerosis
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intrathecal Injection for ALS
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Modifying Protocol
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-7-ATG-7-01
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; ALS; Stem cells
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): three intrathecal injections of 50 million cells at two-month intervals.
  Interventions: Biological: AlloRx

INTERVENTIONS:
Biological: AlloRx — cultured allogeneic adult umbilical cord derived mesenchymal stem cells

SUMMARY:
This trial will study the safety and efficacy of intrathecal injection of cultured allogeneic adult umbilical cord derived mesenchymal stem cells for the treatment of amyotrophic lateral sclerosis

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis is a devastating disease. There is evidence that mesenchymal stem cell treatment is safe and can improve the prognosis of afflicted patients. Patients with ALS will receive three intrathecal injections of cultured allogeneic adult umbilical cord derived mesenchymal stem cells. The dose for each injection will be 50 million cells and the injections will be at two-month intervals. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Amyotrophic Lateral Sclerosis.
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Anticoagulation medicine use
* Clinically significant Abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Previous organ transplant
* Hypersensitivity to sulfur
* Continued drug abuse
* Pre-menopausal women not using contraception

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

SECONDARY OUTCOMES:
Efficacy: revised ALS functional rating scale (ALSFRS-R) | Four year follow-up
  ALSFRS-R scale is used to evaluate the progression of disability in patients with ALS. It will be completed for each follow up point.

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (1):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda

REFERENCES:
- [Background] Cedarbaum JM, Stambler N, Malta E, Fuller C, Hilt D, Thurmond B, Nakanishi A. The ALSFRS-R: a revised ALS functional rating scale that incorporates assessments of respiratory function. BDNF ALS Study Group (Phase III). J Neurol Sci. 1999 Oct 31;169(1-2):13-21. doi: 10.1016/s0022-510x(99)00210-5. PMID 10540002
- [Background] Petrou P, Gothelf Y, Argov Z, Gotkine M, Levy YS, Kassis I, Vaknin-Dembinsky A, Ben-Hur T, Offen D, Abramsky O, Melamed E, Karussis D. Safety and Clinical Effects of Mesenchymal Stem Cells Secreting Neurotrophic Factor Transplantation in Patients With Amyotrophic Lateral Sclerosis: Results of Phase 1/2 and 2a Clinical Trials. JAMA Neurol. 2016 Mar;73(3):337-44. doi: 10.1001/jamaneurol.2015.4321. PMID 26751635
- [Background] Barczewska M, Maksymowicz S, Zdolinska-Malinowska I, Siwek T, Grudniak M. Umbilical Cord Mesenchymal Stem Cells in Amyotrophic Lateral Sclerosis: an Original Study. Stem Cell Rev Rep. 2020 Oct;16(5):922-932. doi: 10.1007/s12015-020-10016-7. PMID 32725316
- [Background] Oh KW, Noh MY, Kwon MS, Kim HY, Oh SI, Park J, Kim HJ, Ki CS, Kim SH. Repeated Intrathecal Mesenchymal Stem Cells for Amyotrophic Lateral Sclerosis. Ann Neurol. 2018 Sep;84(3):361-373. doi: 10.1002/ana.25302. Epub 2018 Aug 31. PMID 30048006